CLINICAL TRIAL: NCT01259232
Title: The Imaging Genetic Study of Schizophrenia and Family
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kunming Medical University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Yuqi Cheng, Kunming Medical University, Kunming Medical University
Other Study IDs: SCH001; KMC2010L4
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- schizophrenia patients,untreated
- schizophrenia relatives
- controls

SUMMARY:
To investigate the brain abnormalities and the association with gene in schizophrenia patients and their relatives.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia（DSM-IV）
* total score of PANSS>64

Exclusion Criteria:

* other psychiatric disease,
* organic disease
* neurological disease
* unstable physiological status
* age>65
* pregnant

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: schizophrenia patients and their relatives
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the association between gene and fMRI in schizophrenia patients | 30 days after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Xu, Study Director — Psychiatry Department
Locations (1):
- Psychiatry department, The 1st Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China